CLINICAL TRIAL: NCT03472625
Title: The Incidence, Severity and Recovery of Aphasia, Dysarthria and Dysphagia Following Stroke in a Tertiary Hospital
Brief Title: The Incidence of Aphasia, Dysarthria and Dysphagia Following Stroke
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201835160
Record Dates: First submitted 2018-03-05; First posted 2018-03-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute stroke patients: All acute stroke patients will be screened for aphasia, dysarthria or dysphagia. When one of the symptoms is present, standardized assessments will follow to evaluate the severity. Recovery in time will be measured +/- 1 week following stroke.
  Interventions: Diagnostic Test: Screening and diagnosis of aphasia, dysarthria, dysphagia

INTERVENTIONS:
Diagnostic Test: Screening and diagnosis of aphasia, dysarthria, dysphagia — Screening (day 2 +/- 1; day 7 +/-1): NIHSS (National Health Institute Scale) 9 and 10 scores, dysphagia screening (nurse), speech-, and language screening (speech therapist)
  Diagnostic assessment (day 2 +/-1-):
  Dysphagia: MASA (Mann Assessment of Swallowing Abilities), FOIS (Functional Oral Intake Scale) Dysarthria: perceptual assessment, NSVO-Z (Nederlands spraakverstaanbaarheidsonderzoek - zinnen) Aphasia: ScreeLing, BNT (Boston Naming Test)

SUMMARY:
The objective of the study is to estimate the incidence and recovery of aphasia, dysarthria and dysphagia in an acute setting (first week) with the NIHSS sub-item scores for language and speech and a dysphagia screening.

Furthermore, we will evaluate the severity of aphasia, dysarthria and dysphagia in an acute setting (first few days) with standardized measurements (ScreeLing, BNT, NSVO-Z, perceptual assessment, MASA/FOIS).

To evaluate the effect of early IVT/EVT in patients with ischemic stroke on functional outcomes for language and speech via the NIHSS scale.

DETAILED DESCRIPTION:
Study population:

Patients who are admitted to the acute Stroke Unit of the University Hospital Ghent will be recruited.

Study course:

The study has a prospective, observational design, with each participant receiving regular standard of care as follows: patients will undergo a clinical examination by a staff neurologists or the present attending in the emergency room. Tailored medical treatment will be given to each patient considering the type of stroke etc. as is standard of care (e.g. thrombolysis and/or thrombectomy for patients with ischemic stroke). Patients that are stable enough are transferred to the Stroke Unit where the neurologist or attending of the unit will reassess all stroke patients. NIHSS scores will be reported at least at day 2 +/- 1. A dysphagia screening is performed by the Stroke Unit nurses when the patient arrives at the Stroke Unit. The scores of the sub-items language and speech of the NIHSS and the dysphagia screening combined with a general screening by a speech language pathologist will be used to confirm or discard aphasia, dysphagia and dysarthria (incidence). When aphasia, dysarthria and/or dysphagia is confirmed, standardized tests will be performed. For this study, data of the following tests will be included for analysis: ScreeLing and/or BNT (aphasia), NSVO-Z and a perceptual assessment (dysarthria), MASA and/or the FOIS (dysphagia). At day 7 +/- 1, NIHSS scores will be reassessed (recovery in time). The diagnostic assessments and the NIHSS sub-items speech/language will be used to investigate the severity and recovery of the symptoms in time. Reports of the neurological clinical examination at follow-up will be retrospectively investigated if possible for additional information about recovery in time.

The total duration of data collection will be approximately 1 week and if possible three months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke patients admitted at the Acute Stroke Unit at the university hospital (Ghent)

Exclusion Criteria:

* Previous aphasia, dysarthria, dysphagia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients recruited at the Acute Stroke Unit (university hospital Ghent)
Sampling Method: Probability Sample
Enrollment: 557 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of aphasia | 3 days
  Incidence is based on the National Institute for Health Stroke Scale (NIHSS), subscale 9. The NIHSS is used to quantify the impairment in patients after stroke. For the incidence of aphasia, subscale 9 of the NIHSS scale is used (best language). It investigates whether a patient has aphasia and what degree if present. Scores on this subscale range from 0 (= normal) to 3 (= mute/global aphasia)

SECONDARY OUTCOMES:
Incidence of dysarthria | 3 days
  based on the National Institute for Health Stroke Scale (NIHSS), subscale 10. This subscale measures whether a patient has dysarthria and if yes, to what degree. Scores range from 0 (= normal) to 2 (= severe dysarthria).
Incidence of dysphagia | 3 days
  based on a nurse screening
Severity of aphasia (screening test) | 3 days
  The severity of aphasia is determined based on a linguistic screening (ScreeLing) performed by a speech pathologist (scores on phonology, semantics, syntaxis)
Severity of aphasia (naming test) | 3 days
  The severity of aphasia is determined based on a naming test (BNT) performed by a speech pathologist
severity of dysarthria (perceptual assessment) | 3 days
  The severity of dysarthria is based on a perceptual assessment performed by the speech pathologist (qualitative assessment)
severity of dysarthria (comprehensibility test) | 3 days
  severity of dysarthria is based on a comprehensibility test (NSVO-Z) performed by a speech pathologist (ranging from 0% to 100% comprehensibility)
severity of dysphagia (swallowing test) | 3 days
  severity of dysphagia is based on a swallowing test (MASA) performed by a speech pathologist
severity of dysphagia (oral intake) | 3 days
  the severity of dysphagia is based on an oral intake scale (FOIS) ranging from 0 (no oral intake) to 7 (normal orale intake)
recovery of aphasia | 1 week, 3 months
  recovery of aphasia is based on the NIHSS 9 at 1 week and 3 months
recovery of dysarthria | 1 week, 3 months
  recovery of dysarthria is based on the NIHSS 10 at 1 week and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: veerle De Herdt, Principal Investigator — University Ghent
Locations (1):
- University Hospital, department of neurology, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Cock E, Batens K, Hemelsoet D, Boon P, Oostra K, De Herdt V. Dysphagia, dysarthria and aphasia following a first acute ischaemic stroke: incidence and associated factors. Eur J Neurol. 2020 Oct;27(10):2014-2021. doi: 10.1111/ene.14385. Epub 2020 Jun 30. PMID 32515514